CLINICAL TRIAL: NCT00232752
Title: A Multicenter, Non-Randomized Study of the 4.0mm Sirolimus-Eluting BX VELOCITYTM Balloon-Expandable Stent in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: Study of the 4.0mm Sirolimus-Eluting Stent in the Treatment of Patients With Coronary Artery Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Mauri Laura, MD, Brigham & Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03-6319
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: 4.0 CYPHER Sirolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: 4.0 CYPHER Sirolimus-Eluting Coronary Stent — 4.0 CYPHER Sirolimus-Eluting Coronary Stent

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the sirolimus-eluting Bx VELOCITYTM stent in reducing in-lesion late loss in patients with de novo native coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female patients minimum 18 years of age
2. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
3. Target lesions treatable with 4mm stent (visual estimate);
4. Target lesion is 30mm in length (visual estimate);
5. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Has unstable angina classified as Braunwald III B or C, or is having a peri infarction;
3. Documented Left ventricular ejection fraction 25%;
4. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2005-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is in-lesion late loss at 6 months post-procedure by QCA. | 6 months post-procedure

SECONDARY OUTCOMES:
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization at 30 days and 6, 9, and 12 months, and 2, 3, 4 and 5 years post-proced | 30 days and 6, 9, and 12 months, and 2, 3, 4 and 5 years post-procedure
Angiographic in-stent and in-lesion binary restenosis (³50% diameter stenosis) 6 months post-procedure by QCA. | 6 months post-procedure
In-stent and in-lesion minimum lesion diameter (MLD) at 6 months post-procedure. | 6 months post-procedure
Target lesion revascularization (TLR) at 6 and 9 months post-procedure. | 6 and 9 months post-procedure
Target vessel revascularization (TVR) at 6 and 9 months post-procedure. | 6 and 9 months post-procedure
Target vessel failure (TVF) at 6 and 9 months post-procedure. | 6 and 9 months post-procedure
Stent lumen and stent obstruction volume by intravascular ultrasound (IVUS) at post-procedure and six months in a subset of approximately 50 patients at selected centers. | post-procedure and six months in a subset of approximately 50 patients
Device success defined as achievement of a final residual diameter stenosis of <50% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used. | End of study
Lesion success defined as the attainment of <50% residual stenosis (by QCA) using any percutaneous method. | End of Study
Procedure success defined as achievement of a final diameter stenosis of <50% (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay. | during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mauri Laura, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States